CLINICAL TRIAL: NCT00279019
Title: A Randomised, Double Blind, Placebo-controlled, Double Dummy, 4-way Cross-over, Dose Ascending Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Inhaled Doses of GSK233705 and Tiotropium Bromide (18µg) Via DPI in COPD Patients
Brief Title: Safety Study Using GSK233705 And Tiotropium In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AC2103473
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK233705; Chronic Obstructive Pulmonary Disease (COPD); COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (16):
- Subjects receiving treatment sequence 1 (Experimental): Eligible subjects will receive treatment sequence 1; GSK233705 20 micrograms, GSK233705 100 micrograms, tiotropium and placebo.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 2 (Experimental): Eligible subjects will receive treatment sequence 2; GSK233705 20 micrograms, Placebo, GSK233705 50 micrograms and tiotropium.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 3 (Experimental): Eligible subjects will receive treatment sequence 3; GSK233705 20 micrograms, tiotropium, Placebo and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 4 (Experimental): Eligible subjects will receive treatment sequence 4; GSK233705 20 micrograms, placebo, tiotropium and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 5 (Experimental): Eligible subjects will receive treatment sequence 5; Placebo, tiotropium, GSK233705 20 micrograms and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 6 (Experimental): Eligible subjects will receive treatment sequence 6; Placebo, GSK233705 20 micrograms, GSK233705 50 micrograms and tiotropium.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 7 (Experimental): Eligible subjects will receive treatment sequence 7; tiotropium, GSK233705 20 micrograms, GSK233705 50 micrograms and Placebo.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 8 (Experimental): Eligible subjects will receive treatment sequence 8; tiotropium, GSK233705 20 micrograms, Placebo and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 9 (Experimental): Eligible subjects will receive treatment sequence 9; GSK233705 20 micrograms, tiotropium, GSK233705 50 micrograms and Placebo.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 10 (Experimental): Eligible subjects will receive treatment sequence 10; GSK233705 20 micrograms, GSK233705 100 micrograms, Placebo and tiotropium.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 11 (Experimental): Eligible subjects will receive treatment sequence 11; Placebo, GSK233705 20 micrograms, tiotropium, and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 12 (Experimental): Eligible subjects will receive treatment sequence 12; Tiotropium, Placebo, GSK233705 20 micrograms and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 13 (Experimental): Eligible subjects will receive treatment sequence 13; Placebo, GSK233705 20 micrograms, GSK233705 50 micrograms and GSK233705 100 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 14 (Experimental): Eligible subjects will receive treatment sequence 14; GSK233705 20 micrograms, placebo, GSK233705 50 micrograms and GSK233705 100 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 15 (Experimental): Eligible subjects will receive treatment sequence 15; GSK233705 20 micrograms, GSK233705 100 micrograms, Placebo and GSK233705 50 micrograms.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo
- Subjects receiving treatment sequence 16 (Experimental): Eligible subjects will receive treatment sequence 16; GSK233705 20 micrograms, GSK233705 100 micrograms, GSK233705 50 micrograms and Placebo.
  Interventions: Drug: GSK233705; Drug: Tiotropium; Drug: Placebo

INTERVENTIONS:
Drug: GSK233705 — GSK233705 will be given orally with dosing strengths of 10, 50, 100 and 250 micrograms/blister via the DISKUS inhaler.
Drug: Tiotropium — Tiotropium will be given orally as overfoiled strips of 5 capsules, each containing 18 micrograms of tiotropium (as bromide monohydrate) administered via a HandiHaler device.
Drug: Placebo — Matching placebo will be given orally as overfoiled strips of 5 capsules, each containing lactose

SUMMARY:
GSK233705 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for once daily treatment of chronic obstructive pulmonary disease (COPD). The long duration of action of GSK233705 when administered via inhalation in animal models supports the potential for use as a once-daily bronchodilator for chronic obstructive pulmonary disease.

GSK233705 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for once daily treatment of chronic obstructive pulmonary disease (COPD). The long duration of action of GSK233705 when administered via inhalation in animal models supports the potential for use as a once-daily bronchodilator for chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion criteria:

* Of non-childbearing potential.
* Diagnosed with COPD, as defined by the GOLD guidelines.
* Smoker or an ex-smoker with a smoking history of at least 10 pack years.
* FEV1/FVC < 0.7 post-bronchodilator (salbutamol).
* FEV1 <= 80% of predicted normal for height, age and gender after inhalation of salbutamol.
* Response to ipratropium bromide 9.
* Subject's weight is 60kg.

Exclusion criteria:

* Past or present disease, which as judged by the Investigator and the Medical Monitor, may affect the outcome of this study.
* FEV1 <=50% of predicted after inhalation of salbutamol.
* Tested positive for hepatitis C antibody, hepatitis B surface antigen or HIV.
* Has claustrophobia that may be aggravated by entering the plethysmography cabinet.
* Has prostate hypertrophy or narrow angle glaucoma.
* Diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, allergic rhinitis, or asthma.
* Poorly controlled COPD.
* Participated in a Pulmonary Rehabilitation Program within 4 weeks prior to screening visit or will enter a program during the study.
* Had a respiratory tract infection in the 4 weeks prior to the screening visit and throughout the duration of the study.
* History of congestive heart failure, coronary insufficiency or cardiac arrhythmia.
* A mean QTc(B) value at screening >440msec, the QTc(B) of all 3 screening ECGs are not within 10% of the mean, a PR interval outside the range 120-210msec or an ECG that is not suitable for QT measurements.
* A history of elevated supine blood pressure or a mean blood pressure equal to or higher than 160/95 mmHg.
* A mean heart rate outside the range 40-90 bpm.
* QTc prolongation >470msec or risk factors for torsades de pointes (heart failure NYHA II-IV, hypokalaemia, familial long QT syndrome).
* Receiving co-medication with drugs which prolong the QTc interval.
* Requires treatment with inhaled cromolyn sodium or nedocromil, oral beta-2-agonists, nebulised beta-2-agonists, nebulised anticholinergics or leukotriene modifiers.
* Unable to abstain from xanthines (other than caffeine.
* Unable to abstain from short-acting inhaled bronchodilators.
* Unable to abstain from long-acting inhaled bronchodilators.
* Changed dose of inhaled or oral corticosteroids within the last 6 weeks.
* Taking more than 10mg/day of prednisolone (or equivalent).
* Receiving treatment with long term or short-term oxygen therapy or requires nocturnal positive pressure for sleep apnea.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-12-12 (Actual); Primary Completion 2006-06-13 (Actual); Study Completion 2006-06-13 (Actual)

PRIMARY OUTCOMES:
Adverse events, blood pressure, heart rate, 12-lead electrocardiogram (ECG), Holter and Lead II ECG monitoring, ECG, lung function and clinical laboratory safety tests. | Up to Week 12

SECONDARY OUTCOMES:
Plasma and urine concentrations of GSK233705 and derived pharmacokinetic parameters. Serial IOS and FEV1 measurements over 27 hours post-dose Serial sGaw, Raw measurements over 24 hours post-dose. | Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours Post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study AC2103473 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/AC2103473?search=study&study_ids=2103473#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC2103473 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register